CLINICAL TRIAL: NCT06304506
Title: Effect of Obesity on Extracellular Matrix Composition in Healthy Males With Normal and High BMI
Brief Title: Effect of Obesity on Extracellular Matrix Composition
Acronym: EOBECM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 514-0894/23-3000
Record Dates: First submitted 2024-02-14; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Adipose Tissue
Keywords: Extracellular matrix compostion; Obesity; Age
MeSH Terms: conditions — Obesity | interventions — Cross-Sectional Studies

STUDY DESIGN:
Intervention Model Description: Cross sectional study with three groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young obese men (Experimental): BMI [30, 40] Age [18, 35]
  Interventions: Other: Cross sectional study
- Young healthy men (Experimental): BMI [20, 25] Age [18, 35]
  Interventions: Other: Cross sectional study
- Old healthy men (Experimental): BMI [20, 25] Age [60, 75]
  Interventions: Other: Cross sectional study

INTERVENTIONS:
Other: Cross sectional study — Physiological testing, Sampling of blood and abdominal adipose tissue and respiratory measurements at rest and during exercise

SUMMARY:
The experiment is a simple cross-sectional study with three groups (n=10) in each group, young and old healthy men and obese young men. The study will investigate the composition of the adipose tissue extra cellular matrix.

The main questions to answer,

- is there differences in the adipose tissue extracellular matrix in obese compared to young men is there differences in the adipose tissue extracellular matrix in old compared to young men

DETAILED DESCRIPTION:
Three groups of young (n=10) and old (n=10) healthy men and obese young (n=10) men are recruited.

After verbal and written information is provided signed consent is obtained.

Subjects arrive at the lab overnight fasted and not having done exercise the prior day and having consumed a normal isocaloric carbohydrate rich diet.

After a voiding and a 15 min rest body composition is determined by DXA. After this blood pressure is measured in the supine position in triplicate separated by 1 min. Following this a venous blood sample is obtained from a cubital vein, and kept on ice until further handling.

Subsequently an adipose tissue biopsy is obtained by the Bergström technique applied with suction from an incision 3-5 cm lateral from the umbilicus. After compression and a 30 min rest, the subject perform an incremental exercise test to determine maximal fat oxidation. In brief pulmonary oxygen uptake and carbon dioxide excretion is measured using a COSMED Quark B2 on-line system during 5 min rest sitting on a cycle ergometer, and then during exercise with 3 min increments starting at 60 Watt and increasing by 35 watts. When the respiratory exchange ratio is above 1 the exercise is stopped. After a 5 min break an incremental test until voluntary exhaustion is performed to determine maximal oxygen uptake. This completes the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged [18,35] and BMI [20,25]
* Obese men aged [18,35] and BMI [30,40]
* Healthy older men aged [60,75] and BMI [20,25]

Exclusion Criteria:

* Present or former cardiovascular disease and chronical inflammatory disease
* Consumption of medications and supplements that influence substrate use at rest and/or during exercise

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The effect of obesity and age on adipose tissue extracellular matrix composition | The human experimental days will be done over the first 6 months of 2024. After informed consent is obtained, each participant will be tested on one day. The laboratory tissue analysis will be performed second half of 2024.
  Adipose tissue extracellular matrix composition will be measured in abdominal subcutaneous adipose tissue sampled 3-5 cm lateral to the umbilicus in 30 male subjects; hereof 10 young, 10 old and 10 young and obese.
  In brief the tissue will be delipidated and subsequently separated by DEAE chromotography (A weak anion exchange) and subsequently analysis of glycosaminoglycan disaccharide composition will be performed by MS.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When the experiments are concluded and the paper(s) are accepted that data will be able upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available after publication and indefinately
Access Criteria: Not known at this state